CLINICAL TRIAL: NCT02117921
Title: Mind Body Syndrome (MBS) Therapy for the Treatment of Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Michael W. Donnino, MA, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000315
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain
Keywords: Mind Body Syndrome; MBS; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- MBS therapy education (Experimental)
  Interventions: Behavioral: One-on-one interview and educational sessions. Reading material for educational series provided.

INTERVENTIONS:
Behavioral: One-on-one interview and educational sessions. Reading material for educational series provided. — A one-on-one interview with the patient and the principal investigator and group educational sessions.

SUMMARY:
To determine if Mind Body Syndrome (MBS) therapy will reduce or eliminate pain in patients suffering from chronic pain syndromes without organic etiology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 18 > years old
* Chronic pain without clear organic etiology after full evaluation by primary care physician or subspecialist
* Pain persistent for a minimum of 3 days a week for the past three months prior to enrollment

Exclusion Criteria:

* Patients < 18 years of age
* Diagnosed organic disease as cause of pain, such as but not limited to malignancy, neurologic disorder (i.e., amyotrophic lateral sclerosis)
* Patients with a diagnosis of significant psychiatric co-morbidities such as schizophrenia and bi-polar disorder. Mild to moderate depression and anxiety will not be considered as exclusions
* Pregnancy
* Severe depression or recent suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory Questionnaire | 4 weeks
  To determine if Mind Body Syndrome (MBS) therapy will reduce or eliminate pain in patients suffering from chronic pain syndromes without organic etiology.
SF-12 Health Survey Scoring Demonstration | 4 weeks

SECONDARY OUTCOMES:
SF-12 Health Survey Scoring Demonstration and Brief Pain Inventory Score | 2 weeks, 4 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No